CLINICAL TRIAL: NCT02092285
Title: Golimumab: A Phase 4, UK, Open Label, Single Arm Study on Its Utilization and Impact in Ulcerative Colitis
Brief Title: Golimumab Utilization and Impact on Ulcerative Colitis (MK-8259-032)
Acronym: GO-COLITIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8259-032; 2013-004583-56 (EudraCT Number)
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golimumab (Experimental): The first induction dose of subcutaneous (SC) golimumab 200 mg was administered at Day 0. The second induction dose of SC golimumab 100 mg was administered two weeks later at Week 2. Responders at Week 6 received a maintenance dose of golimumab (50 mg for participants with a body weight <80 kg or 100 mg for participants with a body weight ≥80 kg) every 4 weeks during the Maintenance Phase for 48 weeks, yielding a total of 54 weeks treatment.
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — 50mg or 100mg solution for injection; subcutaneous injection
  Other Names: Simponi®

SUMMARY:
The primary objective of this study is to evaluate the efficacy of golimumab in maintaining a clinical response in participants with moderate-to-severe ulcerative colitis.

DETAILED DESCRIPTION:
This study consists of a 1 week screening period, a 54 week treatment period, and a 12 week follow-up period, requiring a total of 7 trial site visits: Visit 1(screening visit, Week -1), Visit 2 (enrollment visit, Day 0), Visit 3 (Week 2), Visit 4 (Week 6), Visit 5 (Week 30) and Visit 6 (Week 54) and Visit 7 (follow-up visit, Week 66).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis for at least 3 months with moderate-to-severe disease at enrollment.
* Has a rectal bleeding subscore of 1 or more at baseline.
* No evidence of active, or latent, or inadequately treated infection with Mycobacterium tuberculosis (TB).
* Must be eligible to start golimumab treatment according to the summary of product characteristics.
* Must be naïve to anti-tumor necrosis factor (anti-TNF) therapy.
* Women of childbearing potential or men capable of fathering children must agree to use adequate birth control measures (eg, abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implant, surgical sterilization).
* Women of childbearing potential must test negative for pregnancy at screening.
* Any prior azathioprine / 6-mercaptopurine use was initiated at least 12 weeks prior to enrollment with either stable dosing or discontinued treatment for the 4 weeks immediately prior to enrollment.

Exclusion Criteria:

* Clinical signs of ischaemic colitis, fulminant colitis or toxic megacolon.
* Has evidence of pathogenic bowel infection.
* Has a diagnosis of indeterminate colitis, or clinical findings suggestive of Crohn's disease.
* Has had surgery as a treatment for ulcerative colitis, or is likely to require surgery.
* Has ulcerative colitis which is confined to a proctitis (distal 15 cm or less).
* Has a current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurological disease.
* Has a current immunization with any live virus vaccine or history of immunization with any live virus vaccine within 3 months of baseline.
* Pregnant or lactating, or planning pregnancy while enrolled in the study.
* Has received agents that deplete B or T cells (eg, rituximab or alemtuzumab) within 12 months prior to study inclusion, or continue to manifest depletion of B or T cells more than 12 months after completion of therapy with lymphocyte-depleting agents.
* Has received cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil (MMF) within 8 weeks prior to study inclusion.
* Has used any investigational drugs within 30 days of Screening.
* Has a known hypersensitivity to human immunoglobulin proteins or other components of golimumab.
* Has received methotrexate within 12 weeks prior to enrollment
* Has received rectal corticosteroids or rectal 5-aminosalicylic acid (5-ASA) compounds within 2 weeks prior to enrollment (may be commenced if required after Week 6 in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Merck Sharp & Dohme Ltd., Hoddesdon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Probert CS, Sebastian S, Gaya DR, Hamlin PJ, Gillespie G, Rose A, Tate H, Wheeler C, Irving PM. Golimumab induction and maintenance for moderate to severe ulcerative colitis: results from GO-COLITIS (Golimumab: a Phase 4, UK, open label, single arm study on its utilization and impact in ulcerative Colitis). BMJ Open Gastroenterol. 2018 Jul 7;5(1):e000212. doi: 10.1136/bmjgast-2018-000212. eCollection 2018. PMID 30002864

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 225 participants were screened; 205 participants started treatment after meeting eligibility criteria.
Period: Induction Phase
Arm/Group | Golimumab
Started | 205
Completed | 170
Not Completed | 35
Not completed — Adverse Event | 7
Not completed — Physician Decision | 4
Not completed — Pregnancy | 1
Not completed — Relapse/Recurrence | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 14
Period: Maintenance Phase & Follow-up
Arm/Group | Golimumab
Started | 170
Completed | 60
Not Completed | 110
Not completed — Adverse Event | 22
Not completed — Lost to Follow-up | 1
Not completed — Non-compliance with study drug | 2
Not completed — Physician Decision | 10
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 11
Not completed — Relapse/recurrence | 29
Not completed — Withdrawal by Subject | 11
Not completed — Lack of Efficacy | 23

BASELINE CHARACTERISTICS:
Groups:
- Golimumab: The first induction dose of SC golimumab 200 mg was administered at Day 0. The second induction dose of SC golimumab 100 mg was administered two weeks later at Week 2. Responders at Week 6 received a maintenance dose of golimumab (50 mg for participants with a body weight <80 kg or 100 mg for participants with a body weight ≥80 kg) every 4 weeks during the Maintenance Phase for 48 weeks, yielding a total of 54 weeks treatment.
Arm/Group | Golimumab
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (15.09)
Age, Customized [Number; unit: Participants]
  Adolescents (12-17 years) | 3
  Adults (between 18 and 64 years) | 184
  From 65 to 84 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 123
Partial Mayo Score [Mean (Standard Deviation); unit: Units on a scale] — The Partial Mayo Score (Mayo Score without endoscopy) measures severity of ulcerative colitis. Three sub-scores for stool frequency, rectal bleeding, and physician's global assessment are each graded from 0 to 3 with higher scores indicating more severe disease. Individual sub-scores are then summed to provide the total score ranging from 0 (normal or inactive disease) to 9 (severe disease).
  Units on a scale | 6.4 (1.40)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Partial Mayo Score Response Criteria Through Week 54
Description: The Partial Mayo Score (Mayo Score without endoscopy) measures severity of ulcerative colitis. Three sub-scores for stool frequency, rectal bleeding, and physician's global assessment are each graded from 0 to 3 with higher scores indicating more severe disease. Individual sub-scores are then summed to provide the total score ranging from 0 (normal or inactive disease) to 9 (severe disease). Clinical response is defined as a decrease in PMS of ≥2 points and ≥30% from baseline, plus either a decrease in rectal bleeding subscore of ≥1 point or an absolute rectal bleeding subscore of ≤1. In this outcome measure, the percentage of participants starting treatment at the start of the Induction Phase (Baseline) who obtained clinical response by the end of the Induction Phase (i.e., by Week 6) and maintained clinical response through Week 54 (i.e., had positive clinical responses at both Weeks 30 and 54) are estimated.
Time Frame: Baseline (Week 0), Week 6, Week 30, Week 54
Population: The analysis population for the evaluation of efficacy during the maintenance period was the Full Analysis Set (FAS205) consisting of participants who received at least 1 dose of golimumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Golimumab
Number analyzed (Participants) | 205
Percentage of Participants | 24.9 [19.1 to 31.4]

ADVERSE EVENTS:
Time Frame: Up to 66 weeks
Description: The analysis population for the evaluation of safety was the All Participants as Treated population consisting of any participant who received study medication.
Arm/Group | Golimumab
Serious Adverse Events (participants affected / at risk) | 49/205
Other Adverse Events (participants affected / at risk) | 82/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab (N=205)
BRADYCARDIA (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (2)
CORNEAL EROSION (Eye disorders) | 1 (1)
ULCERATIVE KERATITIS (Eye disorders) | 1 (1)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 (1)
ANAL FISSURE (Gastrointestinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 5 (6)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 23 (23)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
RECTAL FISSURE (Gastrointestinal disorders) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
CLOSTRIDIUM BACTERAEMIA (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 3 (3)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 (2)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MIGRAINE (Nervous system disorders) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab (N=205)
COLITIS (Gastrointestinal disorders) | 15 (15)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 28 (29)
NAUSEA (Gastrointestinal disorders) | 15 (15)
NASOPHARYNGITIS (Infections and infestations) | 20 (22)
HEADACHE (Nervous system disorders) | 15 (18)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to provide to the Sponsor 45 days prior to submission, review copies of abstracts or manuscripts for publication that report any results of the trial. The Sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regards to proprietary information, data accuracy, fairness, and compliance with federal regulations.